CLINICAL TRIAL: NCT07143383
Title: CAMHS and Social Prescribing Applications
Acronym: CASPA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: National Academy for Social Prescribing (Unknown); We Do Wellbeing (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 177012
Record Dates: First submitted 2025-08-19; First posted 2025-08-27 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Mental Health
Keywords: Social prescribing; CAMHS; Mental health; Child; Young person
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Masking Description: Statistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social Prescribing (Experimental): SP is a person-centered approach to wellbeing involving the co-development of a non-clinical prescription, between an individual (i.e. young person) and Link Workers (LWs), based on the perceived difficulties for the referral and the YPs values, needs and preferences. LWs have a good knowledge of their local areas, via community asset mapping and networking, allowing them to connect individuals with different types of available support and activities. Typically, SP ranges from 6-12 sessions (average 8 sessions: unpublished data from sites) with a LW over an 8-week period. Sessions may take place online, via phone call, or in person. As part of this process, LWs draw on psychological skills such as motivational interviewing and behavioral activation as well as employ problem solving and goal setting. Following the identification of issues and preferences, the LW will discuss with the YP what the available local activities and support structures are that match their preferences.
  Interventions: Behavioral: Social Prescribing
- Signposting (Active Comparator): Those in the control group will receive signposting to activities and local sources of support in their communities. This will consist of a CAMHS clinician or researcher meeting with YP identified and providing them with a leaflet detailing the same local sources of support identified by the LW from asset mapping.
  Interventions: Behavioral: Signposting

INTERVENTIONS:
Behavioral: Social Prescribing — SP is a person-centered approach to wellbeing involving the co-development of a non-clinical prescription, between an individual (i.e. young person) and Link Workers (LWs), based on the perceived difficulties for the referral and the YPs values, needs and preferences. LWs have a good knowledge of their local areas, via community asset mapping and networking, allowing them to connect individuals with different types of available support and activities. Typically, SP ranges from 6-12 sessions (average 8 sessions: unpublished data from sites) with a LW over an 8-week period. Sessions may take place online, via phone call, or in person. As part of this process, LWs draw on psychological skills such as motivational interviewing and behavioral activation as well as employ problem solving and goal setting. Following the identification of issues and preferences, the LW will discuss with the YP what the available local activities and support structures are that match their preferences.
  Arms: Social Prescribing
Behavioral: Signposting — Those in the control group will receive signposting to activities and local sources of support in their communities. This will consist of a CAMHS clinician or researcher meeting with YP identified and providing them with a leaflet detailing the same local sources of support identified by the LW from asset mapping.
  Arms: Signposting

SUMMARY:
Background: Social prescribing (SP) is a mechanism for linking patients with non-medical forms of community support and has demonstrated mental health benefits for adults and young people (YP). However, SP is predominantly based in primary care, which limits accessibility for YP who typically engage less with this setting. Within CAMHS (Child and Adolescent Mental Health Services), SP has only recently begun to be trialed, mainly as a pre-treatment option while waiting for care. The CASPA study will pilot a novel SP pathway embedded after the start of psychological treatment in CAMHS, aiming to test its feasibility, acceptability, and potential impact on mental health and wellbeing through a randomized controlled trial.

Methods: CASPA is a two-group (intervention vs. active control) parallel randomized pilot study with YP as the unit of randomization. A total of 120 YP aged 11-18, who have started psychological treatment for emotional difficulties in one of three CAMHS sites in England, will be recruited. Participants in the intervention group will receive a co-produced, person-centered SP pathway involving up to six sessions with a trained Link Worker (LW). These sessions will help identify 'what matters to them' and connect YP with locally mapped community activities and support (e.g. arts, sports, volunteering). Participants in the control group will receive signposting to the same community resources via a leaflet from CAMHS staff or researchers. Quantitative data will be collected at baseline, 3-month and 6-month follow-up, including measures of resilience, mental health, wellbeing, service use, and quality of life. Primary outcomes include feasibility, acceptability, and appropriateness of the intervention, assessed through validated measures and participation metrics, alongside any evidence of impact. Qualitative interviews with YP, CAMHS staff, and LWs will explore implementation experiences, barriers, facilitators, and mechanisms of impact.

Discussion: The CASPA study will generate preliminary evidence regarding the feasibility, acceptability, and appropriateness of offering SP after psychological treatment within CAMHS has started. It will also provide early insights into whether this approach can improve outcomes for YP with emotional difficulties. Findings will inform decisions on the design and justification for a future full-scale clinical and cost-effectiveness trial.

ELIGIBILITY:
Eligibility criteria

Inclusion criteria:

(i) CAMHS

* Wish to participate in CASPA
* Located in England

(ii) YP Participants

* Aged between 11 to 18 years
* Capacity to give assent (if under 16), or
* Capacity to give informed consent (if aged 16 or over or has Gillick competence if aged under 16)
* Have started psychological treatment in CAMHS for an emotional difficulty (e.g. depression, anxiety)

(iii) Parent/Guardian Participants

* Aged 18 or over
* Capacity to give informed consent for YP involvement in CASPA (when the YP is aged between 11-15 and lacks Gillick competence)

(iv) CAMHS staff and LWs:

* Aged 18 or over
* Capacity to give informed consent to participate in CASPA

Exclusion criteria (i) YP participants

• YP with emotional difficulties put on an enhanced specialist pathway due to another severe and complex difficulty which requires intensive input (e.g. anorexia, psychosis or severe and complex difficulties (as judged by the assessing clinician))

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability (young people) | 3 and 6 months
  YP: Acceptability will be assessed using an item from the Friends and Family test, which asks individuals to rate how likely they would be to recommend the service (in this instance, the SP pathway). It is assessed on a five-point Likert Scale, ranging from '1' Extremely Unlikely to '5' Extremely Likely. Higher scores indicate better acceptability.

SECONDARY OUTCOMES:
Acceptability (CAMHS Staff and LWs) | 6 months
  Acceptability of Intervention Measure (AIM) is assessed using 4 questions each on a five-point Likert scale (scoring between 4-20)
Feasibility (young people) | Post intervention (t least 3 months)
  YP will be asked about the feasibility of the intervention via qualitative interviewing where questions can be appropriately framed for their age and experience.
Feasibility (CAMHS Staff and LWs) | 6 months
  Description: Link workers (LW) and CAMHS staff: Feasibility of Intervention Measure (FIM) is assessed using 4 questions each on a five-point Likert scale (scoring between 4-20). Higher scores indicate higher intervention feasibility.
Appropriateness (young people) | 3 and 6 months
  Appropriateness will be assessed by the proportion of sessions offered versus the number the young person attends.
Appropriateness (CAMHS Staff and LWs) | 6 months
  Appropriateness Intervention Appropriateness Measure (IAM) is assessed using 4 questions each on a five-point Likert scale (scoring between 4-20). Higher scores indicate higher intervention appropriateness
Wellbeing: ONS Personal Wellbeing Questions | Baseline, 3 and 6 months
  The Office for National Statistics ONS3 are three subjective measures designed to capture key aspects of personal well-being in the general population. These questions assess three core domains of well-being: evaluative, eudemonic, and affective. Respondents are asked to rate the three questions on a scale from 0 (not at all) to 10 (completely).
  Higher scores reflect greater well-being
Depression: Short Mood and Feelings Questionnaire. | Baseline, 3 and 6 months
  The SMFQ is a 13-item scale questionnaire. Each item reflects core symptoms of depression based on DSM criteria, such as sadness, tiredness, irritability, and feelings of worthlessness. Respondents rate how true each statement has been over the past two weeks on a 3-point Likert scale: "Not True", "Sometimes True", or "True".
  Higher scores reflect greater levels of depressive traits.
Anxiety: Generalised Anxiety Disorder-7 Questionnaire. | Baseline, 3 and 6 months
  The GAD-7 includes 7 items, each reflecting a DSM-IV symptom of generalized anxiety disorder such as excessive worry, nervousness, and difficulty relaxing. Respondents are asked how often they were bothered by each symptom over the past two weeks, using a 4-point Likert scale ranging from "Not at all" to "Nearly every day." Total scores range from 0 to 21, with cutoff points identifying mild (5), moderate (10), and severe (15) anxiety.
Stress: Perceived Stress Scale-4. | Baseline, 3 and 6 months
  The PSS-4 includes four questions evaluating how unpredictable, uncontrollable, and overloaded individuals find their lives. Responses are given on a 5-point Likert scale ranging from 0 ("Never") to 4 ("Very often"). Higher scores indicate greater perceived stress.
Service Use: Short-Client Service Receipt of Inventory. | Baseline, 3 and 6 months
  The CSRI gathers detailed information on service contacts, informal care, medication use, employment, and accommodation over a specified recall period, in this instance, 3 months.
  The first 9 questions on frequency of healthcare service use are scored on a 6-point Likert scale, ranging from 0 'not at all', to 6 'once per day'. Higher scores indicate more contact with services.
  The next 2 questions explore contact with emergency healthcare services (accident and emergency and inpatient admission' and are scored 1 'no' or 2 'yes'. Higher scores indicate more contact with emergency services. For inpatient admission, patients are also asked to specify the number of days they were in hospital.
  The next question explore the impact and support of mental health on an individual's school or workplace. One question asks how many days were missed at school or the individual's workplace because of mental health difficulties. Scores range from 0-93 with higher scores indicating more days missed
Quality of Life: Child Health Utility-9D. | Baseline, 3 and 6 months
  The Child Health Utility-9D (CHU-9D) was developed to address the lack of generic preference-based measures specifically designed for children. The CHU-9D encompasses both shared and unique dimensions compared to other instruments. Common areas include pain and usual activities, while child-specific dimensions include schoolwork/homework, tiredness, and sleep. CHU9D is assessed using 9 questions on a five-point Likert scale (scoring between 1-5). Higher scores indicate higher quality of life.

OTHER OUTCOMES:
Emotional Regulation: ERICA | Baseline, 3 and 6 months
  Mechanism: ERICA is a 17-item tool explicitly developed for youth and designed to assess emotional self-efficacy and regulation strategies in children aged 8 to 16. Its structure covers emotional self-awareness, emotional control, and situational responsiveness, offering a well-rounded view of emotion regulation capacity. Emotional regulation is assessed using 16 questions each on a five-point Likert scale ('1' Strongly disagree to '5' Strongly agree) including 10 questions being reverse scored.
  Higher scores indicate greater emotional regulation.
Community connection: subscale of Student Resilience Survey | Baseline, 3 and 6 months
  Mechanism: using questions from the Student Resilience Survey which is assessed using 4 questions each on a five-point Likert scale (scoring between 4-20). Higher scores indicate higher community connection.
Self-esteem: subscale of Student Resilience Survey | Baseline, 3 and 6 months
  Mechanism: using questions from the Student Resilience Survey which is assessed using 4 questions each on a five-point Likert scale (scoring between 4-20). Higher scores indicate higher self-esteem.
Problem solving: subscale of Student Resilience Survey | Baseline, 3 and 6 months
  Mechanism using the Student Resilience Survey which is assessed using 3 questions each on a five-point Likert scale (scoring between 3-15). Higher scores indicate higher problem solving with others.
Goals and aspirations: subscale of Student Resilience Survey | Baseline, 3 and 6 months
  Mechanism using the Student Resilience Survey which is assessed using 3 questions each on a five-point Likert scale (scoring between 3-15). Higher scores indicate higher levels of goals and aspirations.
Family connection: subscale of Student Resilience Survey | Baseline, 3 and 6 months
  Mechanism: using questions from the Student Resilience Survey which is assessed using 4 questions each on a five-point Likert scale (scoring between 4-20). Higher scores indicate higher family connection.
School connection: subscale of Student Resilience Survey | Baseline, 3 and 6 months
  Mechanism: using questions from the Student Resilience Survey which is assessed using 4 questions each on a five-point Likert scale (scoring between 4-20). Higher scores indicate higher school connection.
Social Structure and Quality. | Baseline, 3 and 6 months
  Mechanism: using questions adapted from PISA 2022 and MCS4 which is assessed using five questions. One of which requires an open-ended numerical value and four questions which are rated on a five-point Likert scale (scoring between 0-16). Higher scores indicate a greater social structure and friendship quality.
Therapeutic Alliance | 3 and 6 months
  Mechanism using the Session Feedback Questionnaire which is assessed using 4 questions each on a five-point Likert scale (scoring between 4-20). Higher scores indicate higher therapeutic alliance. This is for individuals in the social prescribing intervention only.

IPD SHARING:
Plan to Share IPD: Undecided
Some IPD data will be shared but specific data is being currently discussed with the funder. We will update this record when we know more.

REFERENCES:
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Stevens K. Developing a descriptive system for a new preference-based measure of health-related quality of life for children. Qual Life Res. 2009 Oct;18(8):1105-13. doi: 10.1007/s11136-009-9524-9. Epub 2009 Aug 20. PMID 19693703
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] PISA (2022): PISA 2022 Assessment and Analytical Framework. OECD; 2023. doi:10.1787/dfe0bf9c-en
- [Background] ONS (2003). Personal well-being in the UK: April 2022 to March 2023. https://www.ons.gov.uk/peoplepopulationandcommunity/wellbeing/bulletins/measuringnationalwellbeing/april2022tomarch2023
- [Background] MSC (2011): UCL Social Research Institute Centre for Longitudinal Studies (2011). MCS Age 11 Child Self-Completion Questionnaire: England.
- [Background] EBPU. Session Feedback Questionnaire . London; 2012. Available: https://www.corc.uk.net/media/1405/sfq_questionnaire.pdf
- [Background] MacDermott, S. T., Gullone, E., Allen, J. S., King, N. J., & Tonge, B. (2010). The emotion regulation index for children and adolescents (ERICA): A psychometric investigation. Journal of Psychopathology and Behavioral Assessment, 32(3), 301-314. https://doi.org/10.1007/s10862-009-9154-0
- [Background] Demkowicz, O., Panayiotou, M., Ashworth, E., Humphrey, N., & Deighton, J. (2019). The factor structure of the 4-item Perceived Stress Scale in English adolescents. European Journal of Psychological Assessment.
- [Background] Angold, A., Costello, E. J., Messer, S. C., Pickles, A., Winder, F., & Silver, D. (1995). Development of a short questionnaire for use in epidemiological studies of depression in children and adolescents (Vol. 5, pp. 237-249).